CLINICAL TRIAL: NCT02724696
Title: French National Observatory of Patients With Thymic Epithelial Tumor
Acronym: RYTHMIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Other Study IDs: IFCT-1104 RYTHMIC
Record Dates: First submitted 2016-03-22; First posted 2016-03-31 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Thymic Epithelial Tumor
Keywords: Thymic Epithelial Tumor; Cohort study; IFCT
MeSH Terms: conditions — Thymic epithelial tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
RYTHMIC (Réseau tumeurs THYMiques et Cancer) is a French nationwide network for TET with the objective of territorial coverage by regional expert centers and systematic discussion of patients management at national tumor board.

DETAILED DESCRIPTION:
RYTHMIC (Réseau tumeurs THYMiques et Cancer) is a nationwide network for TET appointed in 2012 by the French National Cancer Institute. The objectives of the network are management of clinical tumor boards and central pathologic review of all cases. RYTHMIC Tumor Board is based on initial histopathological diagnosis.

RYTHMIC is a comprehensive tool for research:

* to improve the management of patients
* to monitor dedicated actions
* to screen patients for future translational and clinical trials

ELIGIBILITY:
Inclusion Criteria:

* patient with Thymic Epithelial Tumors

Exclusion Criteria:

* histology other than Thymic Epithelial Tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Thymic Epithelial Tumors
Sampling Method: Non-Probability Sample
Enrollment: 3262 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
histological type | 5 years
  histological type according to the WHO classification 2004/2015
Masaoka-Koga stage | 5 years
  Masaoka-Koga stage
ITMIG/IASLC 2014/2015 stage | 5 years
  ITMIG/IASLC 2014/2015 stage

SECONDARY OUTCOMES:
Questions raised at the national expert multidisciplinary tumor board | 5 years
  Diagnosis/Imaging, Surgery, Chemotherapy, Radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin BESSE, Dr, Principal Investigator — Villejuif - Gustave Roussy
Locations (2):
- France (2):
  - Paris - Institut Curie, Paris
  - Villejuif - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chalabreysse L, Thomas De Montpreville V, De Muret A, Hofman V, Lantuejoul S, Parrens M, Payan MJ, Rouquette I, Secq V, Girard N, Marx A, Besse B, Molina TJ. [Rythmic-pathology: the French national pathology network for thymic epithelial tumours]. Ann Pathol. 2014 Feb;34(1):87-91. doi: 10.1016/j.annpat.2014.01.010. Epub 2014 Feb 21. French. PMID 24630641
- [Result] Hadoux J, Girard N, Besse B. [Thymic epithelial neoplasms: updates on diagnosis, staging, biology and management in France]. Bull Cancer. 2012 Nov;99(11):1045-55. doi: 10.1684/bdc.2012.1659. French. PMID 23131309
- [Result] Thomas de Montpreville V, Quilhot P, Chalabreysse L, De Muret A, Hofman V, Lantuejoul S, Parrens M, Payan MJ, Rouquette I, Secq V, Girard N, Besse B, Marx A, Molina TJ. Glut-1 intensity and pattern of expression in thymic epithelial tumors are predictive of WHO subtypes. Pathol Res Pract. 2015 Dec;211(12):996-1002. doi: 10.1016/j.prp.2015.10.005. Epub 2015 Oct 19. PMID 26534878
- [Result] Remon J, Girard N, Mazieres J, Dansin E, Pichon E, Greillier L, Dubos C, Lindsay CR, Besse B. Sunitinib in patients with advanced thymic malignancies: Cohort from the French RYTHMIC network. Lung Cancer. 2016 Jul;97:99-104. doi: 10.1016/j.lungcan.2016.04.024. Epub 2016 May 3. PMID 27237035
- [Result] Merveilleux du Vignaux C, Dansin E, Mhanna L, Greillier L, Pichon E, Kerjouan M, Clement-Duchene C, Mennecier B, Westeel V, Robert M, Quantin X, Zalcman G, Thiberville L, Lena H, Molina T, Calcagno F, Fournel P, Mazieres J, Besse B, Girard N. Systemic Therapy in Advanced Thymic Epithelial Tumors: Insights from the RYTHMIC Prospective Cohort. J Thorac Oncol. 2018 Nov;13(11):1762-1770. doi: 10.1016/j.jtho.2018.08.005. Epub 2018 Aug 21. PMID 30138763
- [Result] Basse C, Thureau S, Bota S, Dansin E, Thomas PA, Pichon E, Lena H, Massabeau C, Clement-Duchene C, Massard G, Westeel V, Quantin X, Oulkhouir Y, Danhier S, Lerouge D, Tanguy R, Thillays F, Le Pechoux C, Dubray B, Thiberville L, Besse B, Girard N. Multidisciplinary Tumor Board Decision Making for Postoperative Radiotherapy in Thymic Epithelial Tumors: Insights from the RYTHMIC Prospective Cohort. J Thorac Oncol. 2017 Nov;12(11):1715-1722. doi: 10.1016/j.jtho.2017.07.023. Epub 2017 Jul 31. PMID 28774861
- [Result] Drevet G, Collaud S, Tronc F, Girard N, Maury JM. Optimal management of thymic malignancies: current perspectives. Cancer Manag Res. 2019 Jul 22;11:6803-6814. doi: 10.2147/CMAR.S171683. eCollection 2019. PMID 31413632
- [Result] Remon J, Girard N, Mazieres J, Dansin E, Pichon E, Greillier L, Dubos C, Lindsay CR, Besse B. Erratum to "Sunitinib in patients with advanced thymic malignancies: cohort from the French RYTHMIC network" [Lung Cancer, 97 (July 2016), 99-104]. Lung Cancer. 2016 Nov;101:146. doi: 10.1016/j.lungcan.2016.09.014. Epub 2016 Oct 6. No abstract available. PMID 27720478
- [Result] Rouquette I, Taranchon-Clermont E, Gilhodes J, Bluthgen MV, Perallon R, Chalabreysse L, De Muret A, Hofman V, Marx A, Parrens M, Secq V, Thomas de Montpreville V, Galateau-Salle F, Brousset P, Milia J, Girard N, Besse B, Molina TJ, Mazieres J. Immune biomarkers in thymic epithelial tumors: expression patterns, prognostic value and comparison of diagnostic tests for PD-L1. Biomark Res. 2019 Dec 4;7:28. doi: 10.1186/s40364-019-0177-8. eCollection 2019. PMID 31827799
- [Result] Girard N, Merveilleux Du Vignaux C, Molina T, Besse B, Rythmic R. [Thymic tumors]. Rev Prat. 2017 Apr;67(4):430-434. French. PMID 30512890
- [Result] Chalabreysse L, Dubois R, Hofman V, Le Naoures C, Mansuet-Lupo A, de Montpreville VT, De Muret A, Parrens M, Piton N, Rouquette I, Secq V, Singeorzan C, Marx A, Girard N, Besse B, Molina TJ. [Thymoma and squamous thymic carcinoma diagnosis; experience from the RYTHMIC network]. Ann Pathol. 2021 Apr;41(2):154-165. doi: 10.1016/j.annpat.2020.11.002. Epub 2020 Dec 10. French. PMID 33309329
- [Result] Molina TJ, Bluthgen MV, Chalabreysse L, de Montpreville VT, de Muret A, Dubois R, Hofman V, Lantuejoul S, le Naoures C, Mansuet-Lupo A, Parrens M, Piton N, Rouquette I, Secq V, Girard N, Marx A, Besse B. Impact of expert pathologic review of thymic epithelial tumours on diagnosis and management in a real-life setting: A RYTHMIC study. Eur J Cancer. 2021 Jan;143:158-167. doi: 10.1016/j.ejca.2020.11.011. Epub 2020 Dec 11. PMID 33316754
- [Result] Petat A, Dansin E, Calcagno F, Greillier L, Pichon E, Kerjouan M, Clement-Duchene C, Mennecier B, Westeel V, Thillays F, Quantin X, Oulkhouir Y, Thiberville L, Ricordel C, Thomas De Montpreville V, Chalabreysse L, Hofman V, Molina T, Fournel P, Bigay Game L, Besse B, Girard N. Treatment strategies for thymic carcinoma in a real-life setting. Insights from the RYTHMIC network. Eur J Cancer. 2022 Feb;162:118-127. doi: 10.1016/j.ejca.2021.11.028. Epub 2021 Dec 26. PMID 34965496
- [Result] Thomas de Montpreville V, Mansuet-Lupo A, Le Naoures C, Chalabreysse L, De Muret A, Hofman V, Rouquette I, Piton N, Dubois R, Benitez JC, Girard N, Besse B, Marx A, Molina TJ. Micronodular thymic carcinoma with lymphoid hyperplasia: relevance of immunohistochemistry with a small panel of antibodies for diagnosis-a RYTHMIC study. Virchows Arch. 2021 Oct;479(4):741-746. doi: 10.1007/s00428-021-03044-2. Epub 2021 Feb 24. PMID 33629132
- [Result] Benitez JC, Boucher ME, Dansin E, Kerjouan M, Bigay-Game L, Pichon E, Thillays F, Falcoz PE, Lyubimova S, Oulkhouir Y, Calcagno F, Thiberville L, Clement-Duchene C, Westeel V, Missy P, Thomas PA, Maury JM, Molina T, Girard N, Besse B. Central Nervous System Metastases in Thymic Epithelial Tumors: A Brief Report of Real-World Insight From RYTHMIC. J Thorac Oncol. 2021 Dec;16(12):2144-2149. doi: 10.1016/j.jtho.2021.08.008. Epub 2021 Aug 26. PMID 34455064
- [Result] Basse C, Botticella A, Molina TJ, Falcoz PE, Oulkhouir Y, Kerjouan M, Pichon E, Westeel V, Thiberville L, Quantin X, Clement-Duchene C, Khalifa J, Tinier FL, Ginoux M, Thillays F, Mordant P, Besse B, Thomas PA, Pechoux CL, Girard N. RADIORYTHMIC: Phase III, Opened, Randomized Study of Postoperative Radiotherapy Versus Surveillance in Stage IIb/III of Masaoka Koga Thymoma after Complete Surgical Resection. Clin Lung Cancer. 2021 Sep;22(5):469-472. doi: 10.1016/j.cllc.2021.01.020. Epub 2021 Feb 4. PMID 33736940
- [Result] Noel N, Le Roy A, Hot A, Saadoun D, Lazaro E, Levesque H, Le Gouellec N, Meaux-Ruault N, Nguyen T, Costedoat-Chalumeau N, Amieux B, Fontana A, De Gennes C, Fulpin J, Thomas PA, Bluthgen MV, Besse B, Lambotte O. Systemic lupus erythematosus associated with thymoma: A fifteen-year observational study in France. Autoimmun Rev. 2020 Mar;19(3):102464. doi: 10.1016/j.autrev.2020.102464. Epub 2020 Jan 7. PMID 31917264